CLINICAL TRIAL: NCT03774160
Title: Combination HIV Prevention, Linking Prevention and Care, for Hispanic Men
Brief Title: Community and Systems-level HIV Prevention in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01MH109401-04 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-12-12 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Two different districts are being used, one in which the intervention is implemented and the other is a no-intervention comparison site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generacion Actual (Experimental): Generacion Actual includes Community-based and a Health Systems Components. This multi-level intervention reaches out to all MSM/trans by mobilizing them to encourage friends to reduce risk behavior and increase HIV testing, and for HIV+ friends, encourage them to link, stay in care, and take medications regularly. The community based component includes a leadership group, community space, community mobilization events, and group sessions to address a variety of psychosocial issues as well as HIV literacy. The Health Systems component includes sensitization of the HIV testing and care staff to working with MSM and trans, Navigators to help MSM/trans to navigate the complex health system; and positive prevention training of providers; all evidence-based approaches.
  Interventions: Behavioral: Generacion Actual
- Comparison (No Intervention): No intervention is implemented in the comparison arm.

INTERVENTIONS:
Behavioral: Generacion Actual — See description in arm description.
  Other Names: Mpowerment
  Arms: Generacion Actual

SUMMARY:
This project involves adapting 3 new intervention components, and then testing them, in combination with a multi-level, community-based intervention, to promote HIV prevention and sexual health among men who have sex with men and transgender women in Lima, Peru. The total intervention has a community-based intervention and a systems-level intervention at the hospital where people living with HIV get care and medications.

DETAILED DESCRIPTION:
Mpowerment (MP) is an evidence-based community-level, structural, social and behavioral intervention for HIV prevention for young men who have sex with men (MSM). MP targets individual and community empowerment and community mobilization, self-affirmation, sexual self-knowledge and creation of a supportive and affirming social environment. MP has been widely used in the U.S. but not in Peru, with the exception of earlier pilot research. In the earlier research, MP was adapted for the sociocultural issues facing MSM and transgender (trans) women in Peru, and only focused risk reduction and increasing HIV testing. In addition to the MP (which is called the community-based intervention), a health systems component has been added. The health systems includes (1) sensitization of hospital staff (where people living with HIV obtain their medication) to the issues facing transgender women and MSM; (2) the use of Navigators, who help MSM and trans women at the hospital navigate the system of care and remain in care; and (3) a focus on "positive prevention", in which providers talk about the positive aspects of maintaining in care and being virally suppressed instead of only talking about "avoiding death." There is a 2.5 year implementation of the intervention, called "Projecto Orgullo Plus" or Project Pride Plus, which involves a longitudinal cohort of MSM/trans in two large districts of Lima, Peru. Primary outcomes will be unprotected anal sex and HIV testing. Secondary outcomes will be self-reported visits to hospital for care and adherence to medications.

ELIGIBILITY:
Inclusion Criteria:

* Must live in either East Lima District or South Lima District
* identify as man who has sex with men or transgender woman who has sex with men
* be between the ages of 18 - 40

Exclusion Criteria:

* not residing in either East or South District of Lima
* not MSM or transgender woman

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 458 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
condomless anal sex | 37 months post-baseline
  condomless anal sex with HIV+ or unknown status partners, assessed via questionnaire
HIV testing ever | 37 months post-baseline
  if have ever tested for HIV
HIV testing frequency | 37 months post-baseline
  frequency of HIV testing by report on questionnaire

SECONDARY OUTCOMES:
If enrolled in care | 37 months post-baseline
  Has the person, after testing HIV+, enroll in care
Seeking regular HIV care | 37 months post-baseline
  If have seen HIV provider recently by report on questionnaire
Taking medications adherently | 37 months post-baseline
  If have missed any times of taking HIV medications by report on questionnaire
If virally suppressed | 37 months post-baseline
  Has the person been told that he/she is virally suppressed

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Kegeles, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Cayetano Heredia University, Lima, Peru

IPD SHARING:
Plan to Share IPD: No